CLINICAL TRIAL: NCT04455958
Title: A Double-Blind, Randomized, Placebo-Controlled Phase II Study of Lopinavir/Ritonavir Versus Placebo in COVID-19 Positive Patients With Cancer and Immune Suppression in the Last Year
Brief Title: Lopinavir/Ritonavir for the Treatment of COVID-19 Positive Patients With Cancer and Immune Suppression in the Last Year
Status: Withdrawn | Phase: Phase 2 | Type: Interventional
Why Stopped: limited resources
Sponsor: OHSU Knight Cancer Institute (Other)
Collaborators: Oregon Health and Science University (Other)
Responsible Party: Principal Investigator, Jennifer Saultz, Principal Investigator, OHSU Knight Cancer Institute
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: STUDY00021444; NCI-2020-02877 (Registry Identifier: CTRP (Clinical Trial Reporting Program)); STUDY00021444 (Other: OHSU Knight Cancer Institute)
Record Dates: First submitted 2020-07-01; First posted 2020-07-02 (Actual); Last update posted 2021-04-26 (Actual); Status verified 2021-04

CONDITIONS: Hematopoietic and Lymphoid Cell Neoplasm; Malignant Solid Neoplasm; Symptomatic COVID-19 Infection Laboratory-Confirmed
MeSH Terms: conditions — Hematologic Neoplasms | interventions — Lopinavir; lopinavir-ritonavir drug combination

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Group I (lopinavir/ritonavir) (Experimental): Patients receive lopinavir/ritonavir PO BID for 14 days in the absence of disease progression or unacceptable toxicity.
  Interventions: Drug: Lopinavir/Ritonavir; Other: Questionnaire Administration
- Group II (placebo) (Placebo Comparator): Patients receive placebo PO BID for 14 days in the absence of disease progression or unacceptable toxicity.
  Interventions: Drug: Placebo Administration; Other: Questionnaire Administration

INTERVENTIONS:
Drug: Lopinavir/Ritonavir — Given PO
  Other Names: Kaletra
  Arms: Group I (lopinavir/ritonavir)
Drug: Placebo Administration — Given PO
  Arms: Group II (placebo)
Other: Questionnaire Administration — Ancillary studies

SUMMARY:
This phase II trial studies how well lopinavir/ritonavir works in treating COVID-19 positive patients with cancer and a weakened immune system (immune-suppression) in the last year and have mild or moderate symptoms caused by COVID-19. Lopinavir/ritonavir may help to lessen or prevent COVID-19 symptoms from getting worse in cancer patients.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVE:

I. To determine if treatment with lopinavir/ritonavir will decrease progression of symptoms compared to control/placebo.

SECONDARY OBJECTIVES:

I. Determine if treatment improves time to symptom resolution. II. Determine the time to symptom progression. III. Determine time to improvement of participants as defined by complete resolution of symptoms.

IV. Determine the proportion of participants who have severe or critical symptoms and hospital admission.

V. Determine the time to hospital admission for those who develop severe of critical symptoms VI. Determine the proportion of participants with an intensive care unit (ICU) admission.

VII. Determine the proportion of participants receiving ventilator support. VIII. Determine survival of participants enrolled on the study.

EXPLORATORY OBJECTIVES:

I. For patients admitted to the hospital, will determine the following parameters: potassium level, blood oxygen level, creatinine, and blood pressure.

II. Identify obstacles and barriers encountered while implementing a clinical trial in the context of a pandemic caused by a contagious disease and associated social distancing.

OUTLINE: Patients are randomized to 1 of 2 groups.

GROUP I: Patients receive lopinavir/ritonavir orally (PO) twice daily (BID) for 14 days in the absence of disease progression or unacceptable toxicity.

GROUP II: Patients receive placebo PO BID for 14 days in the absence of disease progression or unacceptable toxicity.

After completion of study treatment, patients are followed up 3 times a week until symptoms resolve plus 2 additional weeks thereafter, for up to 3 months, whichever occurs first.

ELIGIBILITY:
Inclusion Criteria:

* Ability to understand and the willingness to sign a written informed consent document
* Participants with a diagnostically proven COVID-19 positive nasal swab test result within 14 days
* Participants must have a diagnosis of cancer
* Participants must be considered immune suppressed either due to their cancer diagnosis or due to treatment of their cancer. Participants must meet at least one of the following criteria:

  * Have received immune suppressing anti-cancer therapy in the past year (i.e., therapy that suppresses white blood cells and/or has been shown to be associated with infection, as stipulated in the drug package insert)
  * Have received intravenous immunoglobulin (IVIG) in the past year for treatment and/or prevention of recurrent infections
  * Are within one year of an autologous bone marrow transplant or chimeric antigen receptor (CAR) T-cell therapy, or within five years of an allogeneic bone marrow transplant
  * Have been treated for three or more infections within the past 6 months
  * Have an absolute neutrophil count at or below 1,500 cells/mcL at some point within two months of the time of consent. This can be due therapy and/or due to cancer suppressing marrow function
  * Have a history of neutropenic fever in the past year
  * Presence of a chronic infection, e.g. tuberculosis (TB) or osteomyelitis, or within 3 months of treatment for such. Topical fungal infections of the skin are not included in this category
* Participants with mild symptoms, must have had mild symptoms for no more than 2 weeks
* Participants with moderate symptoms, must have had moderate symptoms for no more than 1 week
* Pregnant or women of child-bearing potential may be treated if they have no documented lopinavir-associated resistance substitutions
* Aspartate aminotransferase (AST) (serum glutamic-oxaloacetic transaminase [SGOT]) and alanine aminotransferase (ALT) (serum glutamate pyruvate transaminase [SGPT]) =< 3 x upper limit of normal (ULN)
* Total bilirubin =< 2 x ULN (individuals with higher values felt to be consistent with inborn errors of metabolism will be considered on a case-by-case basis)
* Creatinine =< 2 x ULN
* Participants with abnormal blood counts (white blood cell [WBC], platelet, hemoglobin [Hg]) will not be excluded

Exclusion Criteria:

* Participants who do not develop mild to moderate symptoms within 28 days of test results
* Participants with rapid clinical deterioration, in the opinion of the investigator
* Participants experiencing severe symptoms according to COVID-19 Symptom Grading Tool
* History of being human immunodeficiency virus (HIV) positive; by history only; participants do not need to confirm by testing
* Participant has any other concurrent severe and/or uncontrolled medical conditions that would, in the investigator's judgment, may cause unacceptable safety risks, contraindicate patient participation in the clinical study or compromise compliance with the protocol
* Participants receiving any contraindicated medication that in the opinion of the investigator cannot be continued while receiving study drug and cannot be held for the duration of the 14-day study treatment period safely
* History of unstable cardiac disease in the past 6 months
* History of prolonged QT interval, or on other cardiac medications known to prolong the QT interval
* Use of strong inhibitors and inducers of CYP3A4 is prohibited. Lopinavir/ritonavir (L/R) is primarily metabolized by CYP3A4. Therefore, concomitant use of strong inhibitors of CYP3A4 (e.g., ketoconazole, itraconazole, clarithromycin, indinavir, nelfinavir and saquinavir), and inducers of CYP3A (e.g. rifampin, phenytoin, carbamazepine, phenobarbital, St. John's wort) are not permitted. The use of other herbals will be reviewed on a case-by-case basis. If they are deemed to be strong modulators of CYP3A4, patients will be excluded if they are unable or unwilling to stop taking them
* Women who plan to breast feed while on this study are not eligible for participation due to the potential for unnecessary adverse event risks to a child

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2021-05-01 (Estimated); Primary Completion 2021-11-01 (Estimated); Study Completion 2021-11-01 (Estimated)

PRIMARY OUTCOMES:
Severity of symptoms | 3 months
  Will be compared to the time of randomization. The severity of symptoms will be categorized as mild, moderate, severe, or critical according to the grading of symptoms. The proportion of participants with progression to more severe symptoms between treatments groups will be compared using a Fisher's Exact test at a 0.05 significance level.

SECONDARY OUTCOMES:
Clinical benefit rate of lopinavir/ritonavir | 3 months
  Will be defined as improvement on symptoms: yes or no. Will be compared between treatment groups using log-rank test. A 95% confidence interval of treatment rate difference in symptom progression will be calculated by the Wald method.
Time to symptom progression | From randomization to the first documented symptoms progression, assessed up to 3 months
  Will be compared between treatment groups using log-rank test.
Time to improvement of participants | From randomization to first documented complete resolution of symptoms, assessed up to 3 months
  Will be compared between treatment groups using log-rank test.
Time to hospital admission for those who develop severe of critical symptoms | From time of randomization to the time of hospital admission, assessed up to 3 months
  Will be compared between treatment groups using log-rank test.
Intensive care unit (ICU) admission: yes or no | 3 months
  Will be compared using Fisher's exact test, and point and interval estimates will be provided.
Receiving ventilator support: yes or no | 3 months
  Will be compared using Fisher's exact test, and point and interval estimates will be provided.
Overall survival | From randomization to death due to any cause, assessed up to 3 months
  Will be compared using Fisher's exact test, and point and interval estimates will be provided.

OTHER OUTCOMES:
Potassium level | 3 months
  Will be compared between treatments group using t-test or non-parametric comparison if the distribution of lab values are deviated from normal distribution. The proportion of participants of whom lab values are obtained will be tabulated and compared using the chi-square test.
Blood oxygen level | 3 months
  Will be compared between treatments group using t-test or non-parametric comparison if the distribution of lab values are deviated from normal distribution. The proportion of participants of whom lab values are obtained will be tabulated and compared using the chi-square test.
Creatinine level | 3 months
  Will be compared between treatments group using t-test or non-parametric comparison if the distribution of lab values are deviated from normal distribution. The proportion of participants of whom lab values are obtained will be tabulated and compared using the chi-square test.
Blood pressure | 3 months
  Will be compared between treatments group using t-test or non-parametric comparison if the distribution of lab values are deviated from normal distribution. The proportion of participants of whom lab values are obtained will be tabulated and compared using the chi-square test.
Ability to remotely consent, monitor, and treat patients in the context of a pandemic of a contagious disease | 3 months
  Will evaluate on a subjective basis the ability to remotely consent, monitor and treat patients in the context of a pandemic of a contagious disease. The proportion of participants able to be remotely consented, monitored, and treated in the context of a pandemic of a contagious disease will be tabulated and compared using the chi-square test.

CONTACTS AND LOCATIONS:
Overall Officials: Jennifer Saultz, Principal Investigator — OHSU Knight Cancer Institute